CLINICAL TRIAL: NCT04622514
Title: A New Model of Integrated Care of Older Patients With Atrial Fibrillation in Rural China: a Cluster Randomization Trial (the MIRACLE-AF Trial)
Brief Title: New Model of Integrated Care of Older Patients With Atrial Fibrillation in Rural China
Acronym: MIRACLE-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Principal Investigator, Minglong Chen, Deputy Director of the Department of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-SR-027
Record Dates: First submitted 2020-10-18; First posted 2020-11-10 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation; Older; Stroke
Keywords: atrial fibrillation; integrated care; rural China; older; stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment committee members will be blinded to the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Village doctor-led telemedicine integrated care (Experimental): To empower village doctors, a new technology-based model of AF care was established in the intervention group. A digital health support platform was developed by our research team, and a network of teams consisting of village doctors and AF specialists in our research team was established in the intervention group. With the aid of this telemedicine platform, village doctors can receive more support from AF specialists in providing integrated AF care to the rural elderly with AF.
  Interventions: Other: Village doctor-led telemedicine integrated care
- Enhanced usual care (Active Comparator): Usual care plus intensified education to patients, their family members, and their village doctors.
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Other: Village doctor-led telemedicine integrated care — 1. Reorienting the model of care: using of telemedicine platform and online consulting clinic; 2. Coordinating services: contract service by village doctor and on-line AF specialist; 3. Empowering and engaging people: provide village doctor ABC pathway training course; regular visit and drug delivery by village doctor (community support); patients and their family members education.
  Arms: Village doctor-led telemedicine integrated care
Other: Enhanced usual care — 1. Usual care; 2. Intensified education to patients, their family members, and their village doctors.
  Arms: Enhanced usual care

SUMMARY:
This cluster randomization study aims to compare the village-doctor led telemedicine integrated care versus usual care to improve compliance with the Atrial Fibrillation Better Care (ABC) pathway components and outcomes for older patients with atrial fibrillation in rural China.

DETAILED DESCRIPTION:
BACKGROUND Atrial fibrillation（AF) prevalence increases sharply with age, and the risk of stroke, dementia, heart failure and death increases significantly. Integrated care for atrial fibrillation patients using simple ABC pathway ('A' Avoid stroke; 'B' Better symptom management; 'C' Cardiovascular and Comorbidity optimization) is associated with a lower risk of adverse outcomes included all-cause death, composite outcome of stroke/major bleeding/cardiovascular death, and first hospitalization. In China, the prevalence of AF is high, but older people living in rural areas are more vulnerable due to low awareness and treatment gaps caused by various factors. China's rural healthcare system, which is primarily reliant on village doctors, falls short of providing optimal management for AF. To support village doctors in providing integrated care for AF, we have developed a digital health support platform. However, the role of this novel telemedicine-based integrated care for AF patients in rural China remains unclear.

AIM OF THIS STUDY This cluster randomization study aims to compare the village-doctor led telemedicine integrated care versus usual care to improve outcome of older patients with atrial fibrillation in rural China.

DESIGN The MIRACLE-AF China trial is a perspective, cluster randomization clinical trial performed in rural China. We aim to include a minimum of 1000 patients with AF aged 65 years or above from around more than 30 village clinics. Follow-up duration of this study is up to 3 years and all patients are followed up every 3 months by rural doctors. Village clinics will be randomized to either the intervention group (the village-doctor led telemedicine integrated care) or the control group (enhanced usual care).

ELIGIBILITY:
Inclusion Criteria:

1. The village clinics need to be willing and able to provide integrated care to their patients with atrial fibrillation; 2. The village doctors from one village clinic serves all AF patients from 3-5 nearby villages; 3. The village doctors are trained to have a fundamental understanding of telemedicine; 4. Patients are eligible for participation if 1) they are aged 65 years or above; 2) they are diagnosed atrial fibrillation by an ECG, AF specialist, or hospital discharge letter; 3) they agree to receive the medical care provided by village clinics; 4) they provide written informed consent.

-

Exclusion Criteria:

1. Moderate to severe rheumatic mitral stenosis or heart valve replacement history.
2. Presence of ICD or CRT device.
3. Cardiac ablation or surgery <3 months prior to inclusion or being planned.
4. Pulmonary vein isolation or left atrial appendage occlusion history or plan to perform any of the above operations.
5. The life expectancy is less than 1 year.
6. Participation in other clinical trials.

   -

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1039 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome of Stage 1: The proportion of patients who met all the three criteria for the ABC pathway of integrated AF care | 12 months after baseline
  The 'A' criterion referred to stroke prevention or anticoagulation. 'A criterion compliant' implies that either appropriate non-vitamin K antagonist oral anticoagulant (NOACs) use, or warfarin was used with a time in the therapeutic range (TTR) >65%. Patients who were not properly treated with OACs are considered as 'A non-compliant'. The 'B' criterion referred to better symptom control with patient-centered decisions on rate or rhythm control. Patients with an EHRA score of I or II are considered to have good control of AF symptoms ('B compliant'). On the contrary, those with an EHRA score of III or IV were defined as 'B non-compliant', which means their symptoms were insufficiently controlled. The 'C' criterion stands for optimal management of cardiovascular risk factors and other comorbidities. 'C criterion compliant' implies that all the considered risk factors and comorbidities were well controlled or optimally treated. Otherwise, patients were considered as 'C non-compliant'
Primary Outcome of Stage 2: The composite of cardiovascular death, all stroke, worsening of heart failure or acute coronary syndrome, and emergency visits due to AF | 36 months after baseline
  Cardiovascular death was defined as death attributable to myocardial infarction, heart failure, arrhythmia, cardiac perforation or tamponade, or other deaths of cardiac origin. Death caused by ischemic stroke, hemorrhagic stroke, peripheral embolism, and pulmonary embolism was also classified as cardiovascular death. All strokes included ischemic stroke and hemorrhagic stroke. A worsening of heart failure or acute coronary syndrome was defined as the need to be hospitalized or have an emergency visit in conjunction with these conditions

SECONDARY OUTCOMES:
Secondary Outcome of Stage 1: The proportions of patients who meet the criterion for the A component in the ABC pathway | 12 months after baseline
  The 'A' criterion referred to stroke prevention or anticoagulation. Thus, 'A criterion compliant' implies that either appropriate non-vitamin K antagonist oral anticoagulant (NOACs) use, or warfarin was used with a time in the therapeutic range (TTR) >65%. Patients who were not properly treated with OACs are considered as 'A non-compliant'
Secondary Outcome of Stage 1: The proportions of patients who meet the criterion for the B component in the ABC pathway | 12 months after baseline
  The 'B' criterion referred to better symptom control with patient-centered decisions on rate or rhythm control. Patients with an European Heart Rhythm Association (EHRA) score of I or II are considered to have good control of AF symptoms ('B compliant'). On the contrary, those with an EHRA score of III or IV were defined as 'B non-compliant', which means their symptoms were insufficiently controlled
Secondary Outcome of Stage 1: The proportions of patients who meet the criterion for the C component in the ABC pathway | 12 months after baseline
  The 'C' criterion stands for optimal management of cardiovascular risk factors and other comorbidities. 'C criterion compliant' implies that all the considered risk factors and comorbidities were well controlled or optimally treated. Otherwise, patients were considered as 'C non-compliant'
Secondary Outcome of Stage 2: All-cause mortality | 36 months after baseline
  all-cause death
Secondary Outcome of Stage 2: Cardiovascular death | 36 months after baseline
  Cardiovascular death was defined as death attributable to myocardial infarction, heart failure, arrhythmia, cardiac perforation or tamponade, or other deaths of cardiac origin. Death caused by ischemic stroke, hemorrhagic stroke, peripheral embolism, and pulmonary embolism was also classified as cardiovascular death
Secondary Outcome of Stage 2: Ischemic or hemorrhagic Stroke | 36 months after baseline
  All strokes: ischemic or hemorrhagic Stroke
Secondary Outcome of Stage 2: Worsening of heart failure or acute coronary syndrome | 36 months after baseline
  A worsening of heart failure or acute coronary syndrome was defined as the need to be hospitalized or have an emergency visit in conjunction with these conditions
Secondary Outcome of Stage 2: Emergency visit due to AF | 36 months after baseline
  Emergency visit due to AF
Secondary Outcome of Stage 2: Major bleeding | 36 months after baseline
  Major bleeding was defined as fatal bleeding, bleeding in a critical area or organ, or clinically overt bleeding leading to a decrease in the hemoglobin level ≥2 g/dl or transfusion of ≥2 units of packed red cells
Secondary Outcome of Stage 2: Clinically relevant non-major bleeding | 36 months after baseline
  Clinically relevant non-major bleeding referred to bleeding that does not meet the criteria for the ISTH definition of major bleeding but is clinically overt bleeding associated with hospital admission, physician-guided medical or surgical treatment, or a change in antithrombotic therapy.
Secondary Outcome of Stage 2: The proportion of patients who met all the three criteria for the ABC pathway of integrated AF care | 36 months after baseline
  The 'A' criterion referred to stroke prevention or anticoagulation. 'A criterion compliant' implies that either appropriate non-vitamin K antagonist oral anticoagulant (NOACs) use, or warfarin was used with a time in the therapeutic range (TTR) >65%. Patients who were not properly treated with OACs are considered as 'A non-compliant'. The 'B' criterion referred to better symptom control with patient-centered decisions on rate or rhythm control. Patients with an EHRA score of I or II are considered to have good control of AF symptoms ('B compliant'). On the contrary, those with an EHRA score of III or IV were defined as 'B non-compliant', which means their symptoms were insufficiently controlled. The 'C' criterion stands for optimal management of cardiovascular risk factors and other comorbidities. 'C criterion compliant' implies that all the considered risk factors and comorbidities were well controlled or optimally treated. Otherwise, patients were considered as 'C non-compliant'

CONTACTS AND LOCATIONS:
Overall Officials: Minglong Chen, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chu M, Zhang S, Gong J, Yang S, Yang G, Sun X, Wu D, Xia Y, Jiao J, Peng X, Peng Z, Hong L, Wang Z, Li M, Lip GYH, Chen M; MIRACLE-AF Investigators. Telemedicine-based integrated management of atrial fibrillation in village clinics: a cluster randomized trial. Nat Med. 2025 Apr;31(4):1276-1285. doi: 10.1038/s41591-025-03511-2. Epub 2025 Feb 21. PMID 39984634
- [Derived] Li M, Chu M, Shen Y, Zhang S, Yin X, Yang S, Lip GYH, Chen M; MIRACLE-AF Trial Investigators. A Novel Model of Integrated Care of Older Patients With Atrial Fibrillation in Rural China. JACC Asia. 2024 Jul 30;4(10):764-773. doi: 10.1016/j.jacasi.2024.07.006. eCollection 2024 Oct. PMID 39553909